CLINICAL TRIAL: NCT04813926
Title: RiOciguAt UseRs Registry
Brief Title: A Study to Learn About How Well Riociguat Works, How Safe it is and How it is Used Under Real World Conditions in Patients in the United States Who Are Receiving Riociguat for High Blood Pressure in the Arteries That Carry Blood From the Heart to the Lungs (Pulmonary Arterial Hypertension, PAH)
Acronym: ROAR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Xcenda, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21427
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with PAH
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — Follow clinical practice.

SUMMARY:
Pulmonary arterial hypertension (PAH) is a type of high blood pressure in the arteries that carry blood from the heart to the lungs. PAH occurs when the openings in the blood vessels of the lungs get smaller and smaller. These smaller openings can be caused by the following:

* The walls of the arteries tightening
* The walls of the arteries becoming stiff and narrow from an overgrowth of cells The increased pressure in the pulmonary arteries strains the right side of the heart and it begins to fail, causing difficulty breathing and other symptoms. As PAH progresses, symptoms get worse.

There is no cure for PAH, but several medications like endothelin receptor antagonists (ERAs), prostacyclin analogues (PCAs) and riociguat, a soluable guanylate cyclase stimulator, are available to help slow the progression of changes in the pulmonary arteries and help reduce symptoms. Riociguat can be taken together with ERAs and PCAs.

In this study, the researchers want to learn about how well riociguat works, how safe it is when patients take it in 1 of these ways:

* alone
* with ERA
* with PCA
* with ERA and PCA The dosage for each patient will be decided by their doctor. The researchers will review information collected from the patients who have decided with their doctor to start riociguat treatment for their PAH. The study will include about 500 patients in the United States who are at least 18 years old. All of the patients will have either just started taking riociguat or will have been taking it for less than 3 months No investigational products will be administered in this study. Patients will be treated with the Standard of Care (SOC) for PAH. The SOC is the currently appropriate treatment in accordance with scientific evidence and agreed upon in collaboration between medical experts for PAH. There will be no study-mandated visits or treatments.

The patients will be in the study for up to 2 years. During this time, they will visit their doctor every 3 to 6 months as part of the Standard of Care. At these visits, the patients will answer questions about their PAH symptoms and whether they have any medical problems. They will also do exercise tests to see how well they are able to breathe and how tired they get while exercising. The doctors will perform other usual examinations which are part of the Standard of Care such as echocardiograms (images of the heart to show how the heart is working) and a right heart catheters (to measure the pressures in the heart) and will take the usual blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years at the time of riociguat treatment initiation
* Diagnosis of PAH per National Institute for Health and Care Excellence (NICE) 2018 classification
* Decision to initiate treatment with riociguat as per investigator's routine treatment practice made prior to enrollment in the study
* Initiation of riociguat, as per the FDA-approved US label:

  * At enrollment OR
  * ≤90 days prior to enrollment, with a documented titration regimen (defined as all documented dose changes including, but not limited to: starting dose and dates and highest tolerated dose and dates)
* Signed informed consent

Exclusion Criteria:

* Previously treated with and discontinued use of riociguat for any reason prior to study enrollment (discontinuation defined as an interruption of therapy ≥30 days)
* Participating in any of the following:

  1. Blinded clinical trial
  2. Clinical trial involving an unapproved drug
  3. Investigational program with interventions outside of routine clinical practice
* Life expectancy <12 months
* Contraindicated to receive riociguat per the FDA approved US label
* Use of nitrates or NO donors in any form
* Use of PDE5 inhibitors
* PH associated with idiopathic interstitial pneumonias
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US patients aged ≥18 years, diagnosed with PAH, who are naïve to and initiating treatment with riociguat as per the FDA approved US label for PAH - either at study enrollment or have initiated riociguat within 90 days prior to study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
Change of 6-minute walk distance (6MWD) from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
Change of NT-proBNP from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
  NT-proBNP: N-terminal pro-hormone B-type natriuretic peptide
Change of BNP from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
  BNP: B-type natriuretic peptide
Change of clinical PAH scores from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
Change of hemodynamic measurements from RHC from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
  RHC: Right-heart catheterization
Change of ECHO measurements from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
  ECHO: Echocardiogram
Change of laboratory tests from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
Change of NYHA/WHO PH functional class from baseline to Months 6, 12, and 24 | At baseline, Month 6, 12, and 24
  NYHA: New York Heart Association WHO: World Health Organization

SECONDARY OUTCOMES:
Change from baseline to Month 6 and change from baseline to Month 12 in Borg Dysponea Index | At baseline, Month 6 and Month 12
Change from baseline to Month 6 and change from baseline to Month 12 in emPHasis-10 | At baseline, Month 6 and Month 12
Persistence/discontinuation rates for riociguat | Up to 24 months
Reasons for discontinuation of riociguat | At Month 6, 12, and 24 post-baseline
Real-world treatment patterns for riociguat for PAH | Up to 24 months
Demographic of patients treated with riociguat | Up to 24 months
Clinical characteristics of patients treated with riociguat | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (50):
- United States (49):
  - Banner University Medical Center- Phoenix, Phoenix, Arizona
  - Honor Health, Phoenix, Arizona
  - Univ of Arizona College of Medicine, Tucson, Tucson, Arizona
  - UCSF, Fresno, California
  - UC Irvine, Irvine, California
  - Cedar Sinai, Los Angeles, California
  - USC, Los Angeles, California
  - UC Davis, Sacramento, California
  - UCSD, San Diego, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Advent Health, Orlando, Florida
  - Tampa General Hospital USF, Tampa, Florida
  - CCF (Cleveland Clinic Florida), Weston, Florida
  - St Francis Medical Ctr, Columbus, Georgia
  - Northwestern, Chicago, Illinois
  - Loyola, Maywood, Illinois
  - Advocate Christ, Oak Lawn, Illinois
  - KUMC, Kansas City, Kansas
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Mass General, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Beaumont Hospital, Troy, Michigan
  - University of Missouri, Columbia, Missouri
  - St. Louis University, St Louis, Missouri
  - Barnes / Wash U, St Louis, Missouri
  - UNMC, Omaha, Nebraska
  - UNMH, Albuquerque, New Mexico
  - Winthrop, Mineola, New York
  - Northwell Health, New Hyde Park, New York
  - Mount Sinai, New York, New York
  - NYU Langone, New York, New York
  - Columbia, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Integris, Oklahoma City, Oklahoma
  - Legacy Health, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Seton Heart, Austin, Texas
  - UT Southwestern, Dallas, Texas
  - Premier Pulmonary, Denison, Texas
  - Houston Methodist, Houston, Texas
  - Baylor Scott and White, Plano, Texas
  - Richmond Pulmonary Associates, Richmond, Virginia
  - VCU/MCV, Richmond, Virginia
  - Providence, Spokane, Washington
  - Advocate Aurora, Milwaukee, Wisconsin
  - Froedtert/Medical College of Wisconsin, Milwaukee, Wisconsin
- Alliance Pulmonary, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.